CLINICAL TRIAL: NCT02581254
Title: Thin Wire Versus Thick Wire Snare for Cold Snare Polypectomy of Diminutive Polyps- A Randomised Controlled Trial
Brief Title: Thin Wire Versus Thick Wire Snare for Cold Snare Polypectomy of Diminutive Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Eric Lee, Staff Specialist Gastroenterology, Western Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HREC/15/WMEAD/97 (4237)
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Polyps
Keywords: Snare; Polypectomy
MeSH Terms: conditions — Polyps

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thin Wire Snare Arm (Experimental): Use of Thin Wire Snare to resect polyp <10mm
  Interventions: Device: Thin Wire Snare
- Thick Wire Snare Arm (Experimental): Use of Thick Wire Snare to resect polyp <10mm
  Interventions: Device: Thick Wire Snare

INTERVENTIONS:
Device: Thin Wire Snare
  Arms: Thin Wire Snare Arm
Device: Thick Wire Snare
  Arms: Thick Wire Snare Arm

SUMMARY:
Cold snare polypectomy (CSP) is now common practice and has proven to be a safe and effective technique for removal of diminutive polyps. Both thick and thin wire snares are now commonly used for CSP. However, because of their physical characteristics, thick wire snares might leave a higher percentage of residual adenoma at the resection site. Since this may result in a higher risk of recurrence, the technique needs to be optimized. Experts have suggested that a thin wire snare might be more efficient, with a lower risk of residual adenoma at the resection site and consequently a lower risk of recurrence and interval cancer.

DETAILED DESCRIPTION:
Approximately 90% of polyps are smaller than 10 mm. Given the risk of transformation of adenomas into invasive cancer over years, it is important that these adenomas are completely resected.

This will be a double-blind, prospective, randomized controlled trial. All eligible patients referred for a colonoscopy will be able to participate. There will be 2 treatment arms, one arm will be treated with a thin wire snare and the other with a thick wire snare. Patients will be randomised through a computer generated programme and blinded for the type of snare used. The treatment arm will be disclosed to the proceduralist after introduction of the colonoscope into the rectum. After resection of the polyp the defect will be carefully examined by the proceduralist. In case of suspicion of residual adenomatous tissue, a re-excision will be performed. If there's a protrusion noticeable at the resection site, this will be biopsied. Ultimately, the margins of the defect will be biopsied on either side for histological confirmation of complete removal.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to give informed consent to involvement in trial. For patients who do not speak English, an interpreter will be asked to translate the informed consent
* Patients referred to Auburn Hospital Endoscopy Unit for a colonoscopy for whatever reason
* At least 1 lesion <10mm beyond the rectosigmoid junction without any endoscopic features of malignancy
* At least 1 lesion <10mm beyond the rectosigmoid junction that according to the proceduralist, can be safely removed with CSP

Exclusion Criteria:

* Current use of antiplatelets (excluding aspirin) or anticoagulants which have not appropriately been interrupted
* Known coagulopathy
* Pregnancy
* If any doubt about the benign character of the polyp, the patient will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2015-07; Primary Completion 2020-01 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Incomplete resection rate of diminutive polyps | 1 year
  biopsies of the margin are analysed histologically and if any adenoma is found on biopsy, this means the resection with the cold snare was incomplete
Percentage of protrusions | 1 year
  cold snare polypectomy can leave a protrusion in the defect, which has previously been shown to be bunched up submucosa. We will record after every polypectomy if a protrusion was visible and if it depends on the snare whether a protrusion occurs or not

SECONDARY OUTCOMES:
Measurement of the need for second excision in case of endoscopically visual residual adenoma | 1 year
  If there is visible adenoma left after excision, then it is in the patient's best interest that this is resected at the time of the colonoscopy. We record in which cases this was necessary and if it occurred more often with 1 snare type than the other
Post polypectomy bleeding requiring intervention | 1 year
  We will record if there is any rectal bleeding after the colonoscopy and if this required re-intervention to stop the bleeding. We will record if this was more prevalent with 1 snare type.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Dr Lee, FRACP, Principal Investigator — Westmead Hospital
Locations (1):
- Auburn Hosptial, Auburn, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sidhu M, Forbes N, Tate DJ, Desomer L, Lee EYT, Burgess N, van Hattem A, Mcleod D, Cheng E, Cartwright S, Schell A, Hilsden RJ, Heitman SJ, Bourke MJ. A Randomized Controlled Trial of Cold Snare Polypectomy Technique: Technique Matters More Than Snare Wire Diameter. Am J Gastroenterol. 2022 Jan 1;117(1):100. doi: 10.14309/ajg.0000000000001554. PMID 34817440